CLINICAL TRIAL: NCT00344344
Title: A Pilot Study to Evaluate the Efficacy of Refined Methods to Mitigate Indoor Allergens in North Carolina and Boston, Massachusetts Homes
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901016; 01-E-N016
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-09-11

CONDITIONS: Hypersensitivity
Keywords: Asthma; Cockroach; Dust Mite; Extermination; Targeted Cleaning; Allergy; Prevention
MeSH Terms: conditions — Hypersensitivity; Asthma

SUMMARY:
A Pilot Study to Evaluate the Efficacy of Refined Methods to Mitigate Indoor Allergens in North Carolina and Boston, Massachusetts Homes

DETAILED DESCRIPTION:
We propose to conduct a study to evaluate the efficacy of an intensive cockroach and cockroach allergen removal program to mitigate cockroach allergen levels in house dust to less than 8 Units Bla g1 allergen protein per gram vacuumed dust in kitchen and TV/family room samples and less than 2 Units Bla g1 per gram vacuumed dust in bedroom samples. In addition, we propose to test the effectiveness of a method of combined dry steam cleaning in conjunction with Capture (Trademark) carpet cleaning for mitigation of dust mite allergens in bedroom carpeting.

Candidate housing units for cockroach allergen mitigation will be identified through ongoing entomology research projects conducted as part of project NC06405 of the North Carolina Agricultural Research Service, entitled Insect-Specific Target Systems for the Development of Novel Tools for Cockroach Control. This project is directed by Dr. Coby Schal, Department of Entomology at North Carolina State University. Prior to enrollment of homes in the allergen intervention study, up to 10 cockroach infested homes will be sampled only (no intervention) using vacuum and swab sampling procedures described in the intervention study protocol. These visits will be coordinated to coincide with home visits associated with project NC06405 and will not involve intervention or data collection other than dust sample collection. Documentation of cockroach infestations in sampled homes will be accomplished through review of infestation data collected as part of project NC06405 activities. The purpose of these sampling-only visits will be to test and refine sample collection methods, to train study staff on sample collection methodologies, and to confirm the heterogeneity of cockroach allergen distribution within cockroach infested dwellings prior to initiation of the intervention study.

For the intervention study, homes with a past history of cockroach infestation will be contacted. Residents of candidate study homes will be contacted by telephone, provided with a brief overview of the study and interviewed to determine if their home qualifies for participation. The telephone interview will focus on occupant assessments of cockroach infestation levels, history and related topics. Homes that appear to have moderate infestation based on telephone screening information will be scheduled for a Screening Visit. During the Screening Visit, after administration of an informed consent form to a single adult home resident, a home environmental questionnaire will be administered and home environmental observations will be made. In addition, adhesive tape (sticky) traps will be placed for assessment of infestation levels and hand-drawn room layout maps will be constructed documenting sticky trap locations. Approximately 3 days after sticky trap placement, a Baseline visit will be conducted to assess sticky trapping results. If sufficient insects have been trapped, vacuum samples and swab samples will be collected in each of three study rooms for allergen analysis (kitchen, TV/family room, one bedroom. As soon as possible after Baseline sampling is completed, a home will be scheduled for an initial intervention visit, comprised of a general cleaning, occupant education on general principals of integrated pest management. An initial extermination effort will be applied as soon as possible after completion of the general home cleaning and an initial targeted cleaning, focused on areas of high allergen concentration as determined by swab sampling results, will occur within 10-15 days of the extermination. At 1, 2, and 4 month points after the initial targeting cleaning, sticky trapping will be performed to confirm the effectiveness of the extermination, both vacuum and swab sampling will be repeated, a brief occupant follow-up questions will be administered and occupant education will be enforced. Based upon the results of sticky trappings, extermination efforts may be repeated. Targeted cleaning will be conducted if any follow-up swab or vacuum samples contain detectable Bla g1 allergen. Six month follow-up visits will also be conducted and will be identical to the 1, 2 and 4 month visits except that they will not include repeated extermination, targeted cleaning activities or occupant education. Recruitment will continue until 16 homes have been enrolled into the cockroach intervention arm of the study, with a goal of completion of at least 12 homes in North Carolina through 6 month follow-up visit. Up to 5 multi-unit dwellings will be enrolled from the inner city Boston, Massachusetts area in order to test this mitigation strategy in inner-city, multiunit dwellings in the Northeastern U.S.

Candidate dust mite intervention homes will be recruited through local advertisements and person to person communication to identify and enroll 8 homes with bedroom carpet dust that contains combined levels of Der f1 and Der p1 of > 10 ug/gram vacuumed dust. Intervention will be applied in a single bedroom and will consist of installation of impermeable bedding covers, occupant education, and carpet steam cleaning followed by Capture (Trademark) cleaning of carpeting. Follow-up vacuumed dust sampling will occur at 1, 2, 4, and 6 month time points and will be immediately followed by repeated steam cleaning followed by Capture (trademark) cleaning at the 1, 2, and 4 month time points. Completion of 6 homes through the 6 month follow-up visit is projected. Only local North Carolina homes will be enrolled into the dust mite allergen intervention.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for the study, each home must:

1. have a home occupant who intends to live at the same address for at least 6 months;
2. have a home occupant live at the house full time;
3. have a home occupant that is at least 21 years of age;
4. have at least one bedroom with wall to wall carpeting.
5. Yield dust collected during the screening visit that contains combined Der f I plus Der p I allergen levels of greater than or equal to 10 ug/gram dust.

   For the intervention arm only:
6. home occupant must have an adult at home during the study visits on weekdays over the six month period that the study is ongoing.

EXCLUSION CRITERIA:

Homes will be excluded from this study if any of the inclusion criteria are not met.

Indoor Dust Mite Allergen:

Must have a home occupant who intends to live at the same address for at least 6 months; live at the house full time; be at least 21 years of age; have at least one bedroom with wall to wall carpeting; yield dust collected during the screening visit that contains combined Def fl plus Der pl allergen levels of greater than or equal to 10 ug/gram dust.

For Intervention arm only - home occupant must have an adult at home during the study visits on weekdays over the six month period that the study is ongoing.

Indoor Cockroach Allergen:

Must have a home occupant that intends to live at the same address for at least 6 months; live in the house full time; be at least 21 years of age; have moderate to severe cockroach infestation as evidenced by occupant self-reports of cockroach sightings and by sticky trap assessment that yield a combined total sticky trap count of 50-250 cockroaches.

For intervention arm only - home occupant must have an adult at home during most of the weekdays over the six month period that the study is ongoing.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88
Dates: Start 2000-10-19; Study Completion 2006-09-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Environmental Health Sciences (NIEHS), Bethesda, Maryland, United States